CLINICAL TRIAL: NCT07011472
Title: ACE Pilot 3: Decision Aid 2 Options vs 3 Options
Brief Title: Post-Operative Analgesic Selection in Patients Planned for Third Molar Extraction After Undergoing Shared Decision Making Using 2- Versus 3-Option Decision-Aids
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Cecile A. Feldman, DMD, Dean, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro2025000930
Record Dates: First submitted 2025-05-21; First posted 2025-06-08 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Pain Management; Shared Decision Making
Keywords: Analgesic selection; shared decision making; decision aid; non-opioid analgesic
MeSH Terms: conditions — Agnosia | interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Decision-Aid with 2-options (Active Comparator): Participants in this arm will undergo a shared decision making process using a decision aid that offers 2 options for post-operative analgesic: a non-opioid combination (ibuprofen/acetaminophen) or an opioid (hydrocodone). Subsequently, their choice for post-operative analgesic will be recorded.
  Interventions: Other: Decision-Aid with 2-options
- Decision-Aid with 3-options (Active Comparator): Participants in this arm will undergo a shared decision making process using a decision aid that offers 3 options for post-operative analgesic: [1] a non-opioid combination (ibuprofen/acetaminophen), [2] an opioid (hydrocodone), or [3] a non-opioid combination plus an opioid prescription for "just-in-case" pain management. Subsequently, their choice for post-operative analgesic will be recorded.
  Interventions: Other: Decision aid with 3 options

INTERVENTIONS:
Other: Decision-Aid with 2-options — This decision aid offers 2 options for post-operative analgesic: a non-opioid combination (ibuprofen/acetaminophen) or an opioid (hydrocodone).
  Arms: Decision-Aid with 2-options
Other: Decision aid with 3 options — This decision aid offers 3 options for post-operative analgesic: a non-opioid combination (ibuprofen/acetaminophen), an opioid (hydrocodone), or a non-opioid combination with a "just-in-case" opioid prescription.
  Arms: Decision-Aid with 3-options

SUMMARY:
This research protocol is exploring a behavioral intervention: shared decision making with the use of a decision aid to select a post-operative analgesic. Specifically, the investigators will examine the impact of shared decision making on analgesic selection for acute pain management when 2 options are presented to the patient as compared to 3 options which includes an opioid prescription for "just-in-case" pain management. The investigators hypothesize that significantly more patients will choice an opioid option when the "just-in-case option is included.

DETAILED DESCRIPTION:
Dentists often prescribe opioids to their patients to manage acute post-surgical pain, with hydrocodone/acetaminophen being the most commonly prescribed opioid combination. With an estimated 56 million tablets of hydrocodone prescribed to 3.5 million high school and young adults each year after third molar extractions, it is vitally important to develop the best evidence for acute pain management following dental procedures.

Dentists are among the leading prescribers of opioid analgesics, writing up to 12% of all opioid prescriptions and 31% of opioid prescriptions for young patients. Shared decision making is an integral component of patient-centered clinical care. Decision aids have been shown to be effective in improving patient satisfaction, and one study suggests shared decisions have the potential to decrease the number of opioids tablets prescribed. Shared decision making studies on analgesics selection for out-patient surgery, however, are limited and no studies have investigated the "just in case" phenomenon which send a message that the opioid options are better than the non-opioid options.

ELIGIBILITY:
Inclusion Criteria:

* Be able to understand the informed consent.
* Provide signed and dated informed consent form
* Be able to understand all directions for data gathering instruments in English
* Be willing and able to comply with all study procedures
* Planning to undergo extraction of one or more 3rd molars
* Be 18 years or older

Exclusion Criteria:

While the actual analgesic prescribed to the patient may be different then the analgesic selected by the participant (their actual analgesic is NOT part of the research protocol) participants who self-report inability to take ibuprofen, acetaminophen or an opioid are not eligible since the decision aid is designed to help a patient select between a combination of ibuprofen/acetaminophen and an opioid containing analgesic.

Participants would also be excluded due to any additional criteria that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study which includes:

* Prior participation in this study
* Inability or refusal to provide informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
% participants selecting opioid analgesics versus non-opioid analgesics | Day 1
  •To determine difference in proportion of patients who choose an opioid option for analgesics after participation in a shared decision making process using a decision aid

CONTACTS AND LOCATIONS:
Locations (1):
- Rutgers School of Dental Medicine, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No